CLINICAL TRIAL: NCT01675297
Title: For 12months, the Multi Center, Randomized, Open-label, Active Controlled Comparative Clinical Study to Assess the Efficacy and the Safety of Risedronate, Cholecalciferol Combination Tablet in Patients With Osteoporosis
Brief Title: Efficacy and Safety Study of Risedronate, Cholecalciferol Combination Tablet in Patients With Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL_RSNP_401
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis
Keywords: Risedronate, cholecalciferol, BMD
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risendronate/Cholecalciferol combination (Experimental): Risendronate/Cholecalciferol combination Risenex Plus tablet: one tablet once a week for 12months
  Interventions: Drug: Risedronate/Cholecalciferol combination
- Risedronate (Active Comparator): Sedron tablet: one tablet once a week for 12months
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate/Cholecalciferol combination — Risendronate/Cholecalciferol combination once a week
  Other Names: RisenexPlus tablet
  Arms: Risendronate/Cholecalciferol combination
Drug: Risedronate — Risedronate once a week
  Other Names: Sedron 35mg tablet
  Arms: Risedronate

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of Risedronate, cholecalciferol combination tablet in patients with Osteoporosis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and the safety of Risedronate with and without cholecalciferol on vitamin D status, Bone Mineral Density (BMD) and bone markers.

ELIGIBILITY:
Inclusion Criteria:

1. Male osteoporosis patients over 19 years of age
2. Female osteoporosis patients with menopause

   * Definition of osteoporosis

     * They had a BMD T-score -2.5 or less at mean Lumbar spine(L1-L4), Femoral neck or total. Or evidence of at least one vertebral fracture
   * Definition of menopause(can be one of three condition)

     * For 12months spontaneous amenorrhea
     * For 6months spontaneous amenorrhea with serum FSH(Follicle stimulating hormone) is 40mlU/mL and over
     * 6weeks after bilateral ovariectomy whether hysterectomy or not.

Exclusion Criteria:

1. Patients with esophagus disorder (i.e:esophagostenosis)
2. Patients administered with osteoporosis therapy(except calcium, Vit.D medication)within the previous 3 Months
3. Patients with serum calcium concentrations 8.0mg under
4. Patients with severe nephropathy (CCr 30mL/min less)
5. Patients with unable to sit upright or stand for 30minutes

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2011-07-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Moo Park, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-ang university hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Pre-assignment Details: wash out 7~14days
Groups:
- Risendronate/Cholecalciferol Combination: Experimental: Administer Risendronate/Cholecalciferol combination one tablet once a week for 12months.
  Risedronate/Cholecalciferol combination: once a week
- Risedronate: Active comparator: Administer Risendronate one tablet once a week for 12months.
  Risedronate: once a week
Period: Overall Study
Arm/Group | Risendronate/Cholecalciferol Combination | Risedronate
Started | 806 | 247
Completed | 642 | 199
Not Completed | 164 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risendronate/Cholecalciferol Combination | Risedronate | Total
Number analyzed (Participants) | 806 | 247 | 1053
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.77 (7.87) | 65.51 (8.59) | 65.71 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 754 | 236 | 990
  Male | 52 | 11 | 63
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.40 (3.32) | 23.00 (3.00) | 23.31 (3.25)
Osteoporosis disease period [Mean (Standard Deviation); unit: years] | 23.90 (37.49) | 27.07 (40.44) | 24.65 (38.21)

OUTCOME MEASURES:

1. Primary Outcome: The Change of Bone Mineral Density (BMD) Value
Description: Higher Bone Mineral Density(BMD) value mean a better outcome.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Risendronate/Cholecalciferol Combination | Risedronate
Number analyzed (Participants) | 642 | 199
g/cm^2
  baseline | 0.77 (0.11) | 0.77 (0.10)
  12 months | 0.81 (0.12) | 0.80 (0.11)
  change(12months-baseline) | 0.04 (0.05) | 0.03 (0.04)

2. Secondary Outcome: The Change of 25OHD(25-hydroxyvitamin D)
Description: range of 25OHD: 4.80~52.80 Higher 25OHD scores mean a better outcome.
  If there is missing data, LOCF(Last Observation Carried Forward) was applied and analyzed.
Time Frame: baseline, 6months, 12months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Risendronate/Cholecalciferol Combination | Risedronate
Number analyzed (Participants) | 642 | 199
ng/ml
  25OHD(baseline) | 18.23 (11.59) | 17.83 (10.99)
  25OHD(6months) | 28.93 (11.16) | 19.47 (12.53)
  25OHD(12months) | 30.57 (11.89) | 18.35 (11.73)
  25OHD change(6months-baseline) | 10.74 (11.53) | 1.68 (9.47)
  25OHD change(12months-baseline) | 12.33 (13.33) | 0.53 (12.74)

3. Secondary Outcome: PTH(Parathyroid Hormone Value)
Description: range of PTH: 13~54 Higher PTH scores mean a worse outcome.
  If there is missing data, LOCF(Last Observation Carried Forward) was applied and analyzed.
Time Frame: baseline, 6months, 12months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Risendronate/Cholecalciferol Combination | Risedronate
Number analyzed (Participants) | 642 | 199
pg/ml
  PTH(baseline) | 40.48 (30.95) | 39.17 (34.04)
  PTH(6months) | 37.34 (23.82) | 42.40 (27.79)
  PTH(12months) | 39.17 (19.37) | 45.27 (23.68)
  PTH change(6months-baseline) | -2.78 (23.36) | 3.39 (35.57)
  PTH change(12months-baseline) | -1.34 (27.31) | 6.16 (33.33)

ADVERSE EVENTS:
Time Frame: 12months
Description: The safety evaluation was conducted in the safety set(Risendronate/Cholecalciferol Combination: 806, Risendronate: 247) Safety set means exclude do not administering investigational product.
Arm/Group | Risendronate/Cholecalciferol Combination | Risedronate
All-Cause Mortality (participants affected / at risk) | 9/806 | 1/247
Serious Adverse Events (participants affected / at risk) | 61/806 | 19/247
Other Adverse Events (participants affected / at risk) | 61/806 | 29/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risendronate/Cholecalciferol Combination (N=806) | Risedronate (N=247)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elderly (Social circumstances) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risendronate/Cholecalciferol Combination (N=806) | Risedronate (N=247)
Dyspepsia (Gastrointestinal disorders) | 20 (21) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (5)
Nasopharyngitis (Infections and infestations) | 19 (22) | 8 (9)

LIMITATIONS AND CAVEATS:
Multiple centers proceded clinical study do not use the same measuring instrument.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes